CLINICAL TRIAL: NCT03287869
Title: A Multicenter, Open-label Trial to Evaluate the Safety and Tolerability of Brexpiprazole in the Treatment of Subjects With Bipolar I Disorder
Brief Title: A Trial to Evaluate the Safety and Tolerability of Brexpiprazole in the Treatment of Participants With Bipolar I Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 331-201-00083; 2017-002225-38 (EudraCT Number)
Record Dates: First submitted 2017-08-24; First posted 2017-09-19 (Actual); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Bipolar I Disorder; Acute Mania
Keywords: Bipolar; Mania; Brexpiprazole
MeSH Terms: conditions — Mania | interventions — brexpiprazole

STUDY DESIGN:
Intervention Model Description: Group composed of eligible rollover participants who completed one of the double-blind, phase 3 efficacy trials (331-201-00080 (NCT03259555) or 331-201-00081 (NCT03257865)).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brexpiprazole (Experimental): Brexpiprazole was administered in participants orally with flexible dosing from 2 mg/day from Days 1 to 3 regardless of treatment assignment in the previous double-blind trial, followed by titration to 3 mg/day on Day 4. Participants may have been titrated (or re-titrated) to a higher dose of brexpiprazole, up to a maximum of 4 mg/day, based on treatment response and at the investigator's discretion anytime at Day 7 or thereafter. Participants who were unable to tolerate their current dose could have been titrated down to a minimum of 2 mg/day any time after Day 4.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole tablets
  Other Names: OPC-34712

SUMMARY:
This study evaluated the safety and evaluate the safety and tolerability of open-label brexpiprazole (2 - 4 mg/day, with a starting dose of 2 mg/day) for the treatment of adult subjects with bipolar I disorder. All participants received a starting dose of brexpiprazole.

DETAILED DESCRIPTION:
While the availability of atypical antipsychotics had increased the therapeutic options available, there remains a need for safer and more effective therapies in the treatment of manic and depressive episodes of bipolar I disorder. Brexpiprazole's specific receptor activity profile likely correlates with its established efficacy in schizophrenia and major depressive disorder, and may prove to be an effective target for the treatment of acute mania of bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria (rollover participants from 331-201-00080 & 331-201-00081 trials)

* Participants remaining in hospital at the Day 21 visit of trial 331-201-00080 or 331-201-00081 were permitted to enroll in the 331-201-00083 trial at the week 3 visit of the double-blind trial if they were planned to be discharged from the hospital before the week 1 visit of trial 331-201-0083. Participants not discharged by the week 1 visit of trial 331-201-0083 were withdrawn.
* Participants who, in the opinion of the investigator, could potentially benefit from administration of oral brexpiprazole for the treatment of bipolar I disorder and who completed 3 weeks of post-randomization treatment in Trial 331-201-00080 & Trial 331-201-00081.

Exclusion Criteria (rollover participants from 331-201-00080 & 331-201-00081 trials)

* Participants with a major protocol violation during the course of their participation in the double-blind phase 3 trials (331-201-00080 or 331-201-00081).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (44):
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - Citrials Inc., Bellflower, California
  - Radiant Research, Cerritos, California
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Apostle Clinical Trials, Long Beach, California
  - Pacific Research Partners, LLC, Oakland, California
  - NRC Research Institute, Orange, California
  - Asclepes Research Centers, PC, Panorama City, California
  - CI Trials, Riverside, California
  - CNRI-San Diego, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - CI Trials, Santa Ana, California
  - Collaborative Neuroscience Network, LLC, Torrance, California
  - Shreenath Clinical Service, Yorba Linda, California
  - Optimus U Corp, Coral Gables, Florida
  - Segal Trials, Fort Lauderdale, Florida
  - Galiz Research, Hialeah, Florida
  - Research Centers of America, LLC, Hollywood, Florida
  - Florida Behavioral Medicine, Largo, Florida
  - University of South Florida Board of Trustees, Tampa, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - NeuroPsychiatric Research, Winfield, Illinois
  - Louisiana Clinical Research, Shreveport, Louisiana
  - CBH Health, Gaithersburg, Maryland
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Arch Clinical Trials, LLC, St Louis, Missouri
  - St. Louis Clinical Trials, St Louis, Missouri
  - Hassman Research Institute, LLC, Berlin, New Jersey
  - Clinical Trials of America-NC, LLC, Hickory, North Carolina
  - Richard H Weisler, MD PA Associates, Raleigh, North Carolina
  - SP Research PLLC, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Pillar Clinical Research LLC, Garland, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
  - Core Clinical Research, Everett, Washington
  - Mid Columbia Research, Richland, Washington
- Bulgaria (9):
  - Mental Health Center Prof. Dr. Ivan Temkov - Burgas EOOD, Department for Treatment of Emergency Psychiatric Condition, Burgas
  - State Psychiatry Hospital - Kardzhali,Third Male Department, First Female Department, Kardzhali
  - State Psychiatry Hospital Sv. Ivan Rilski, First Male department, First Female Department, Novi Iskar
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Clinic of Psychiatry, Plovdiv
  - "Mental Health Centre-Ruse" EOOD, Male department for persons with severe mental disorders, Female department for persons with severe mental disorders, Rousse
  - University Multiprofile Hospital for Active Treatment -Alexandrovska EAD, Clinic of Psychiatry, First Department of Psychiatry, Sofia
  - Multiprofile Hospital for Active Treatment - Targovishte AD, Department of Psychiatry, Targovishte
  - Mental Health Center - Veliko Tarnovo EOOD, Department of Psychiatry for Active Treatment of Persons with Severe Mental Disorders, Veliko Tarnovo
  - Mental Health Center - Vratsa EOOD, Department of Psychiatry, Vratsa
- Croatia (2):
  - CHC Rijeka-Clinic for Psychiatrics, Rijeka
  - Poliklinika Neuron /Polyclinic Neuron, Zagreb
- Poland (2):
  - Indywidualna Specjalistyczna Praktyka Lekarska Wieslaw Jerzy Cubala, Gdansk
  - NZOZ Prywatna Klinika Psychiatryczna Inventiva, Tuszyn
- Serbia (6):
  - CHC Dr Dragisa Misovic, Belgrade
  - Clinic for Psychiatric Disorders, Dr Laza Lazarevic, Belgrade
  - Clinic for Psychiatry, Belgrade
  - Specialized Hospital for Psychiatry Diseases Kovin, Kovin
  - Clinical Center Kragujevac, Clinic of Psychiatry, Kragujevac
  - Klinika za psihijariju, Klinicki Centar Vojvodine, Novi Sad
- Ukraine (10):
  - Regional Clinical Hospital n.a I.I. Mechnicov, Dnipro
  - SI of Neurology Psychiatry and Narcology NAMS, Kharkiv
  - Kherson Regional Psychiatric Hospital, Kherson
  - Kyiv Regional Medical Incorporation Psychiatry, Kyiv
  - CI of LOR Lviv Regional Clinical Psychiatric Hospital, Department #25, Lviv
  - Communal Institution of Lviv Regional Council "Lviv Regional Clinical Psychiatric Hospital", department #20, Lviv
  - Odesa Regional Psychiatric Hospital 2, Odesa
  - Maltsev Regional Clinical Psychiatric Hospital, Poltava
  - Ternopil Regional Municipal Clinical Psychoneurological Hospital, Ternopil
  - O.I. Yushenko Vinnitsa Regional Clinic, Vinnitsa

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included participants who completed 3-week double-blind treatment in studies 331-201-00080 (NCT03259555)/331-201-00081 (NCT03257865) and, who in the investigator's judgment, could potentially benefit to receive brexpiprazole in this study. Data was summarized as per the treatment received in the previous studies.
Groups:
- Prior Brexpiprazole: Brexpiprazole was administered in participants orally with flexible dosing from 2 mg/day from Days 1 to 3 regardless of treatment assignment in the previous double-blind trial, followed by titration to 3 mg/day on Day 4. Participants may have been titrated (or re-titrated) to a higher dose of brexpiprazole, up to a maximum of 4 mg/day, based on treatment response and at the investigator's discretion anytime at Day 7 or thereafter. Participants who were unable to tolerate their current dose could have been titrated down to a minimum of 2 mg/day any time after Day 4. Participants who received brexpiprazole in the double-blind treatment period in previous studies were included in this group.
- Prior Placebo: Brexpiprazole was administered in participants orally with flexible dosing from 2 mg/day from Days 1 to 3 regardless of treatment assignment in the previous double-blind trial, followed by titration to 3 mg/day on Day 4. Participants may have been titrated (or re-titrated) to a higher dose of brexpiprazole, up to a maximum of 4 mg/day, based on treatment response and at the investigator's discretion anytime at Day 7 or thereafter. Participants who were unable to tolerate their current dose could have been titrated down to a minimum of 2 mg/day any time after Day 4. Participants who received placebo in the double-blind treatment period in previous studies were included in this group.
Period: Overall Study
Arm/Group | Prior Brexpiprazole | Prior Placebo
Started | 188 | 193
Analyzed For Safety (Safety Sample) (Participants who received at least 1 dose of investigational medicinal product (IMP-brexpiprazole).) | 184 | 184
Completed | 105 | 100
Not Completed | 83 | 93
Not completed — Adverse Event | 14 | 12
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 13 | 19
Not completed — Non-Compliance With Study Drug | 5 | 9
Not completed — Progressive Disease | 1 | 0
Not completed — Protocol Deviation | 2 | 1
Not completed — Withdrawal by Subject | 36 | 43
Not completed — Early Closure of the Site | 0 | 1
Not completed — Physician Decision | 5 | 5
Not completed — Reason not Specified | 6 | 3

BASELINE CHARACTERISTICS:
Population: Enrolled Sample included all participants who signed an inform consent form (ICF) for the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prior Brexpiprazole | Prior Placebo | Total
Number analyzed (Participants) | 188 | 193 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (11.0) | 46.1 (11.5) | 45.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 92 | 189
  Male | 91 | 101 | 192
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 129 | 146 | 275
  Race: Black or African American | 52 | 47 | 99
  Race: American Indian or Alaska Native | 3 | 0 | 3
  Race: Asian | 2 | 0 | 2
  Race: Race-Other | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 21 | 24 | 45
  Ethnicity: Not Hispanic or Latino | 165 | 169 | 334
  Ethnicity: Ethnicity-Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event (TEAE) by Severity
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. AEs severity were graded on a 3-point scale as: 1 = mild; discomfort noticed, but no disruption to daily activity, 2 = moderate; discomfort sufficient to reduce or affect normal daily activity, and 3 = severe; inability to work or perform normal daily activity.
Time Frame: From Day 1 (after dosing) through 29 weeks (26 weeks treatment, 3 weeks safety follow-up)
Population: Safety Sample included all participants who received at least 1 dose of IMP (brexpiprazole).
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 184 | 184
Participants
  TEAE, Any grade | 79 | 86
  TEAE, Mild | 60 | 68
  TEAE, Moderate | 31 | 29
  TEAE, Severe | 8 | 5

ADVERSE EVENTS:
Time Frame: From Day 1 (after dosing) through 29 weeks (26 weeks treatment, 3 weeks safety follow-up)
Description: Safety Sample included all participants who received at least 1 dose of IMP.
Arm/Group | Prior Brexpiprazole | Prior Placebo
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/184
Serious Adverse Events (participants affected / at risk) | 11/184 | 8/184
Other Adverse Events (participants affected / at risk) | 13/184 | 26/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prior Brexpiprazole (N=184) | Prior Placebo (N=184)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 2 (2)
Mania (Psychiatric disorders) | 5 (5) | 1 (1)
Suicidal Behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prior Brexpiprazole (N=184) | Prior Placebo (N=184)
Akathisia (Nervous system disorders) | 8 (9) | 17 (17)
Headache (Nervous system disorders) | 5 (5) | 10 (12)

LIMITATIONS AND CAVEATS:
As predefined in the protocol, there were no primary or secondary efficacy endpoints in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03287869/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT03287869/SAP_003.pdf